CLINICAL TRIAL: NCT04709237
Title: Evaluation of The Clinical Acceptance of Soft Contact Lenses for Myopia Control
Status: Completed | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-20-51
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Results first posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2022-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | Unapproved Device: Yes

ARMS (3):
- Omafilcon A Control Lens first, then Omafilcon A Test Lens 1, then Omafilcon A Test Lens 2 (Experimental): Participants wore three different types of study contact lenses (1 control and 2 test contact lenses), in a randomized order of testing for the three study contact lens types.
  Interventions: Device: omafilcon A control lens; Device: omafilcon A test lens 1; Device: omafilcon A test lens 2
- Omafilcon A Test Lens 2 first, then Omafilcon A Control Lens , then Omafilcon A Test Lens 1 (Experimental): Participants wore three different types of study contact lenses (1 control and 2 test contact lenses), in a randomized order of testing for the three study contact lens types.
  Interventions: Device: omafilcon A control lens; Device: omafilcon A test lens 1; Device: omafilcon A test lens 2
- Omafilcon A Test Lens 1 first, then Omafilcon A Control Lens , then Omafilcon A Test Lens 2 (Experimental): Participants wore three different types of study contact lenses (1 control and 2 test contact lenses), in a randomized order of testing for the three study contact lens types.
  Interventions: Device: omafilcon A control lens; Device: omafilcon A test lens 1; Device: omafilcon A test lens 2

INTERVENTIONS:
Device: omafilcon A control lens — Participants were randomized to wear omafilcon A control soft contact lens for 10 days.
Device: omafilcon A test lens 1 — Participants were randomized to wear omafilcon A test soft contact lens 1 for 10 days.
Device: omafilcon A test lens 2 — Participants were randomized to wear omafilcon A test soft contact lens 2 for 10 days.

SUMMARY:
The main objective of the study was to evaluate the clinical acceptance of soft contact lenses for Myopia control.

DETAILED DESCRIPTION:
Participants were randomized to wear each study contact lenses for 10 days with investigator and participant masking. The participants who are not contact lens wearer at enrollment wore single vision contact lenses for two weeks during the pre-investigation phase to get adapted to contact lens wear.

ELIGIBILITY:
Inclusion Criteria:

* Age 10 to 16 years;
* Spectacle refraction: -0.75 to -6.00D spherical equivalent, maximum anisometropia 1.25D, cylinder up to -1.00DC
* Best corrected visual acuity of at least 20/25 in each eye.
* Parents/guardians and participant have read and understood the Participant Information Sheet;
* Parents/guardians and participant have read, signed and dated the Informed Consent;
* Have normal eyes with the exception of the need for visual correction;
* Be willing and able to adhere to the instructions set in the clinical protocol and maintain the appointment schedule.

Exclusion Criteria:

* Ocular anterior segment infection, inflammation, abnormality, or active disease that would contraindicate contact lens wear;
* Newly prescribed use of some systemic or ocular medications for which contact lens wear could be contraindicated as determined by the investigator;
* Monocular participants (only one eye with functional vision) or participants fit with only one lens;
* Subjects with slit lamp findings greater than grade 1 (e.g. edema, infiltrates, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival, anterior segment inflammation) as per ISO 11980, any previous history or signs of a contact lens related corneal inflammatory event (past corneal ulcers), or any other ocular abnormality that may contraindicate contact lens wear at the enrolment visit;
* History of herpetic keratitis, ocular surgery or irregular cornea;
* Enrolment of the family members of the investigator, family members of the investigator's staff, or individuals living in the households of these individuals.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2019-12-14 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ocular Technology Group - International, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Omafilcon A Control Lens First, Then Omafilcon A Test Lens 1, Then Omafilcon A Test Lens 2: Participants first wore omafilcon A control lens first, followed by the other 2 study contact lenses in a randomized order. Each study lens was worn for 10 days.
- Omafilcon A Test Lens 2 First, Then Omafilcon A Control Lens , Then Omafilcon A Test Lens 1: Participants first wore omafilcon A test lens 1, followed by the other 2 study contact lenses in a randomized order. Each study lens was worn for 10 days.
- Omafilcon A Test Lens 1 First, Then Omafilcon A Control Lens , Then Omafilcon A Test Lens 2: Participants first wore omafilcon A test lens 2, followed by the other 2 study contact lenses in a randomized order. Each study lens was worn for 10 days.
Period: Overall Study
Arm/Group | Omafilcon A Control Lens First, Then Omafilcon A Test Lens 1, Then Omafilcon A Test Lens 2 | Omafilcon A Test Lens 2 First, Then Omafilcon A Control Lens , Then Omafilcon A Test Lens 1 | Omafilcon A Test Lens 1 First, Then Omafilcon A Control Lens , Then Omafilcon A Test Lens 2
Started | 7 | 7 | 7
Completed | 6 | 7 | 7
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Nineteen total participants were analyzed out of the 20 participants who completed the study. One participant was not included in the analysis because of the compliance issue (Did not complete required hours with lens).
Groups:
- Overall Study: Nineteen total participants were analyzed out of the 20 participants who completed the study.
Arm/Group | Overall Study
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.4 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Overall Vision Satisfaction
Description: Overall vision satisfaction recorded on a visual analog scale of 0 to100 (0 - Not Happy, 100 - Very Happy)
Time Frame: 10 days
Population: 19 total participants were analyzed out of the 20 participants. One participant was not included in the study because of the compliance issue (Did not complete required hours with lens).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Omafilcon A Control Lens: Participants wore omafilcon A Control Lens during the study.
- Omafilcon A Test Lens 1: Participants wore omafilcon A Test Lens 1 during the study.
- Omafilcon A Test Lens 2: Participants wore omafilcon A Test Lens 2 during the study.
Arm/Group | Omafilcon A Control Lens | Omafilcon A Test Lens 1 | Omafilcon A Test Lens 2
Number analyzed (Participants) | 19 | 19 | 19
units on a scale | 87.7 (12.1) | 79.7 (16.5) | 71.8 (27.3)

2. Primary Outcome: Habitual Daily Wearing Time
Description: Habitual daily wearing time in hours
Time Frame: 10 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours/Day
Arm/Group | Omafilcon A Control Lens | Omafilcon A Test Lens 1 | Omafilcon A Test Lens 2
Number analyzed (Participants) | 19 | 19 | 19
Hours/Day | 7.9 (2.0) | 8.1 (2.2) | 7.8 (2.3)

3. Secondary Outcome: Visual Acuity
Description: Visual acuity measured using logMAR
Time Frame: 10 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Omafilcon A Control Lens | Omafilcon A Test Lens 1 | Omafilcon A Test Lens 2
Number analyzed (Participants) | 19 | 19 | 19
logMAR | 0.06 (0.07) | 0.08 (0.07) | 0.10 (0.09)

4. Secondary Outcome: Overall Visual Satisfaction During the Use of iPad With White Screen
Description: Visual satisfaction during specific visual tasks on visual analog scale of 0 to100 (0 - Not Happy, 100 - Very Happy)
Time Frame: 10 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A Control Lens | Omafilcon A Test Lens 1 | Omafilcon A Test Lens 2
Number analyzed (Participants) | 19 | 19 | 19
units on a scale | 90.8 (9.3) | 90.8 (10.0) | 85.1 (16.2)

5. Secondary Outcome: Visual Satisfaction During the Use of Ipad With White Screen- How Clear is the Close-up Vision.
Description: Visual satisfaction during specific visual tasks on visual analog scale of 0 to100 (0 - Not Clear at All, 100 - Very Clear)
Time Frame: 10 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A Control Lens | Omafilcon A Test Lens 1 | Omafilcon A Test Lens 2
Number analyzed (Participants) | 19 | 19 | 19
units on a scale | 90.7 (9.5) | 90.0 (13.3) | 84.4 (15.4)

6. Secondary Outcome: Visual Satisfaction During the Use of iPad With Black Screen- How Happy the Vision is.
Description: Visual satisfaction during specific visual tasks on visual analog scale of 0 to100 (0 - Not Happy, 100 - Very Happy)
Time Frame: 10 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A Control Lens | Omafilcon A Test Lens 1 | Omafilcon A Test Lens 2
Number analyzed (Participants) | 19 | 19 | 19
units on a scale | 85.4 (16.1) | 86.8 (15.7) | 80.0 (20.0)

7. Secondary Outcome: Visual Satisfaction During the Use of Ipad With Black Screen- How Clear is the Close-up the Vision is.
Description: as for outcome 5
Time Frame: 10 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A Control Lens | Omafilcon A Test Lens 1 | Omafilcon A Test Lens 2
Number analyzed (Participants) | 19 | 19 | 19
units on a scale | 85.3 (14.0) | 87.5 (15.1) | 79.2 (22.3)

ADVERSE EVENTS:
Time Frame: Duration of all three study lens wear for approximately 30 days.
Arm/Group | Omafilcon A Control Lens | Omafilcon A Test Lens 1 | Omafilcon A Test Lens 2
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 2/19 | 0/19 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omafilcon A Control Lens (N=19) | Omafilcon A Test Lens 1 (N=19) | Omafilcon A Test Lens 2 (N=19)
Headache (Product Issues) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omafilcon A Control Lens (N=19) | Omafilcon A Test Lens 1 (N=19) | Omafilcon A Test Lens 2 (N=19)
Headache (General disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT04709237/Prot_SAP_001.pdf